CLINICAL TRIAL: NCT06792461
Title: A Randomized Controlled Trial to Evaluate the Implementation of an eHealth Platform for Promoting Healthy Habits Among Adolescents From Socially Disadvantaged Settings: the ePro-Schools Project
Brief Title: ePlatform for Promoting Health in Schools
Acronym: ePro-Schools
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Universitat Autonoma de Barcelona (Other); Parc Sanitari Sant Joan de Déu (Other); Universitat Oberta de Catalunya (Other); Consorcio Centro Investigación Biomédica en RED (CIBER)-SAM (Unknown); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Utrecht University (Other); Klaipėda University (Other); Technical University of Munich (Other); Riga Stradins University (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Rodrigo Antunes Lima, Researcher, Fundació Sant Joan de Déu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24/099-P; 101095426 (Other Grant/Funding Number: ERA4Health)
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Health Promotion; Health Education; Physical Activity; Nutrition; Behaviour Change
Keywords: eHealth; Adolescents; Socially disadvantaged settings; Randomized control trial; Co-design; School-based interventions; Health promotion
MeSH Terms: conditions — Health Education; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Schools will be randomized to one of the two groups and all students, their families, teachers and other school staff within those schools will be placed in the respective group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants (students, parents, teachers, and other school staff) will have access to a series of resources and training with the ultimate goal of promoting healthy lifestyles among adolescents. This material will be delivered via the ePro-Schools platform throughout one school year (2025/26). This platform will be available in web-based format and contents will be provided through two formats: the intervention platform (with content for teachers and students) and the information platform (with content for teachers, students, and families).
  Interventions: Behavioral: Physical activity and nutritional behavioural intervention
- Control group (No Intervention): Participants in the control group will have access to the information platform, which will contain basic information about health-related habits (healthy eating and physical activity) during the 2025/26 school year. Participants in the control group will have access to the intervention platform after the completion of the trial.

INTERVENTIONS:
Behavioral: Physical activity and nutritional behavioural intervention — The ePro-Schools intervention includes two digital platforms designed to promote physical activity and healthy nutrition among adolescents:
  1. The Intervention Platform, which provides interactive content for both students and PE teachers.
  2. The Information Platform, which offers educational resources for students, teachers, and families.
  The intervention content-currently being refined through a co-creation process-will feature engaging modules focused on physical activity and healthy eating. Adolescents will have access to more than 15 interactive modules, while PE teachers will benefit from 8 targeted pedagogical modules aimed at enhancing their lessons and encouraging greater student participation in physical activity.
  Control group will have access to the information platform
  Arms: Intervention group

SUMMARY:
There are few public health and educational policies specifically aimed at promoting physical activity, healthy dietary habits, and reducing sedentary behaviour among adolescents from socially disadvantaged backgrounds. ePro-Schools will co-design, pilot and evaluate an evidence-based program, delivered via a modular eHealth platform, to promote physical activity and healthy eating, and reduce time in sedentary behaviours. A profound co-creation process involving adolescents, school staff, and policymakers-alongside the adaptation of previous interventions by consortium members-will support the program's development. The ePro-Schools platform will contain modules for adolescents and their parents, teachers and school administration. Although the platform will be implemented through schools, it will include content to be implemented outside the school setting. The intervention program will be evaluated through a randomised controlled trial conducted in six secondary schools in Central Catalonia that aims to include 1000 adolescents. Schools have been randomised (1:1) into an intervention and a waiting-list control group.

The evaluation of the program includes effectiveness, cost-effectiveness and process evaluation. Physical activity, sedentary behaviour and eating habits are the primary effectiveness outcomes of the trial. Secondary outcomes include fitness, water consumption, quality of life, depressive symptoms, social isolation and sleep quality. Using implementation science methodology, ePro-Schools will co-design transferable evidence-based practices and methodologies and guidance for scaling up the platform with policymakers and stakeholders, as well as informing specialists, policymakers and the general public.

DETAILED DESCRIPTION:
There is limited high-quality information regarding physical activity, sedentary behaviour and dietary habits focusing on adolescents from socially disadvantaged settings. Therefore, there is a limited number of public health and educational policies specifically designed for this population group. The ePro-Schools project will address both knowledge gaps in the state-of the-art by co-designing and testing the effectiveness of an intervention, which includes an eHealth platform (website), for promoting healthy habits among adolescents from socially disadvantaged settings in the area of Central Catalonia. For this reason, the main aim of the ePro-Schools project is to co-design and test the effectiveness of an eHealth platform for promoting healthy habits among adolescents from socially disadvantaged settings. The specific objectives of the project are to:

1. Co-design with adolescents and teachers from secondary schools and policymakers in socially disadvantaged settings a modular and digital eHealth platform for promoting healthy habits among adolescents.
2. Pilot test with adolescents and teachers from secondary schools the ePro-Schools platform
3. Conduct a randomized controlled trial (RCT) in a group of schools located in socially disadvantaged settings in Catalonia to evaluate the effectiveness, cost-effectiveness and implementation parameters of the ePro-Schools program in regard to physical activity, sedentary behaviour and dietary habits of adolescents in socially disadvantaged settings.
4. Evaluate to which extend changes in lifestyle behaviours (physical activity, sedentary behaviour and dietary habits) are associated with physical and mental health in adolescents from socially disadvantaged settings.
5. Co-design with adolescents, teachers and policymakers transferable evidence-based practices, methodologies and guidance for upscaling of the ePro-Schools platform as a public mental health policy for youth, and present it to EU, national and regional policymaker.

The study will be conducted in the area of Central Catalonia, particularly in six secondary schools from socially disadvantaged settings (intervention group vs control group size ratio 1:1). We will focus on students attending 1st, 2nd and 3rd year of secondary school, and in total, around 1000 adolescents will be involved. Moreover, physical activity teachers and school staff from the selected secondary schools will participate in the study as well. The families of the adolescents will also be involved in the study.

To achieve all the objectives, the project has several phases:

1. Co-design (Objective 1): The platform will be co-created with input from various stakeholders-adolescents, teachers, school administrators, and policymakers. Focus group sessions with teachers and school directors will shape the content and features of the platform, while policymakers will provide feedback on potential barriers and strategies for large-scale implementation.
2. Project Survey (Objective 1): A survey will be conducted with teachers and students to gather feedback on the platform's content, particularly regarding physical activity and nutrition.
3. Pilot Testing (Objective 2): After the co-creation phase, alpha and beta testing of the platform will occur, including feedback from stakeholders and experts. A pilot test will assess usability, functionality, and integration of feedback to refine the platform before the main trial.
4. Randomized Controlled Trial and Evaluation (Objectives 3 & 4): In a randomized controlled trial, control group will receive basic health-related information, while the intervention group will use the ePro-Schools platform. Participants will be evaluated at multiple time points to assess the impact on lifestyle behaviors, physical health, and mental well-being.
5. Co-design of Transferable Practices (Objective 5): A concluding workshop with stakeholders will consolidate findings and generate actionable recommendations for scaling the platform, resulting in a policy translation report to guide broader implementation.

The RCT will be evaluated regarding its effectiveness, cost-effectiveness and process implementation.

Regarding the effectiveness of the program, statistical analyses will assess the impact of the program using Mixed Methods with Repeated Measurements (MMRM) for continuous data and Generalized Estimating Equations (GEE) for categorical data. The analyses will measure outcomes at both post-intervention and follow-up, adjusting for potential confounders (e.g., sex, sociodemographic status, and baseline outcomes). For the cost-effectiveness, a comparison of costs between the new intervention and regular care will be made, calculating the incremental cost-effectiveness ratio (ICER). The cost-effectiveness will be expressed as cost per Quality-Adjusted Life Year (QALY) gained. The implementation evaluation will focus on evaluating the adoption, acceptability, appropriateness, and feasibility of the program. Adoption will be assessed through multiple indicators, such as questionnaire completion and content interaction, instead of just logins or time spent on the platform. Acceptability and feasibility will be evaluated using questionnaires, interviews, and focus groups during the co-creation phase. Barriers and facilitators to intervention implementation will also be explored.

ELIGIBILITY:
Inclusion Criteria

Adolescents:

* Students enrolled in 1st, 2nd, or 3rd year of ESO (ages approximately 11-16) at participating secondary schools located in the Central Catalonia region, particularly those in socially disadvantaged settings.
* All genders will be eligible.
* Written informed consent must be provided by both the adolescent and their parent(s)/legal guardian(s).

Physical Education Teachers:

* Physical education teachers currently working at the participating secondary schools.
* Must be 18 years of age or older.
* Must provide written informed consent to participate.

Exclusion Criteria

* Individuals (adolescents or teachers) who do not provide written informed consent will be excluded.
* No other exclusion criteria will be applied.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Physical activity level | Participants will be evaluated at baseline (pre-intervention), at the end of the school year (post-intervention) and at follow-up (nine months after post-intervention)
  The level of physical activity will be measured with the PAQ-A questionnaire. It consists of 10 questions that assess different aspects of physical activity levels, using a 5-point Likert scale, although only 9 questions are used to calculate the final score.
Physical activity intensities | Participants will be evaluated at baseline (pre-intervention), at the end of the school year (post-intervention) and at follow-up (nine months after post-intervention)
  The intensity of physical activity will be measured with the IPAQ questionnaire. It consists of a series of questions that assess three different intensities of physical activity: light, moderate and vigorous.
Sedentary behaviour | Participants will be evaluated at baseline (pre-intervention), at the end of the school year (post-intervention) and at follow-up (nine months after post-intervention)
  Sedentary behaviour will be measured with the IPAQ questionnaire using the question regarding sedentary behaviour (time spent in sedentary behaviours)
Dietary habits | Participants will be evaluated at baseline (pre-intervention), at the end of the school year (post-intervention) and at follow-up (nine months after post-intervention)
  Dietary habits and food consumption that will be assessed by PREDIMED test. This test is based on Mediterranean Diet items regarding healthy eating habits. It is composed by 13 questions. The PREDIMED score will be calculated as follow: <9 points (classified as low adherence) and >9 (classified as high adherence). The higher the score, the healthier the adolescent food habits are.

SECONDARY OUTCOMES:
Child Health Utility | Participants will be evaluated at baseline (pre-intervention), at the end of the school year (post-intervention) and at follow-up (nine months after post-intervention)
  Quality of life which will be assessed by Child Health Utility 9D Index. It is a paediatric generic preference-based measure of health-related quality of life. The questionnaire has 9 questions with 5 response levels per question.
  Scoring: Each participant's responses define a unique health state, which is converted into a single utility score ranging from 0 (equivalent to being dead) to 1 (full health) considering their country and age group.
Physical fitness | Participants will be evaluated at baseline (pre-intervention), at the end of the school year (post-intervention) and at follow-up (nine months after post-intervention)
  The physical fitness assessed by the European physical fitness test: Eurofit. It is a standardized set of physical and functional tests designed to assess physical fitness. Teachers will report the students' results since this is a test already implemented in the school. The tests performed are: Cardiorespiratory endurance (20-meter endurance shuttle run), Muscle Strength (standing broad jump), Speed (30m sprint), and Agility (shuttle run: 10 x 5m).
Water consumption | Participants will be evaluated at baseline (pre-intervention), at the end of the school year (post-intervention) and at follow-up (nine months after post-intervention)
  Participants will be asked how many glasses of water they drink per day.
Well-being | Participants will be evaluated at baseline (pre-intervention), at the end of the school year (post-intervention) and at follow-up (nine months after post-intervention)
  Well-being assessed by the Kidscreen-10 test. The questionnaire use 5-point Likert-type scales to assess either the frequency (never-seldom-sometimes-often-always) of certain behaviors/feelings or, in a smaller number of cases, the intensity of an attitude (not at all-slightly moderately very-extremely).
  The Kidscreen-10 test measures quality of life in 10 dimensions: Physical Well-Being, Psychological Well-Being, Moods and Emotions, SelfPerception, Autonomy, Relations with Parents and Home Life, Social Support and Peers, School Environment, Social Acceptance (Bullying) and Financial Resources.
  Scoring: The scores for the 10 items are summed to produce a total score between 10 and 50 points, where the higher the score, the higher the wellbeing.
Depressive symptomatology | Participants will be evaluated at baseline (pre-intervention), at the end of the school year (post-intervention) and at follow-up (nine months after post-intervention)
  Depressive symptomatology assessed by the Center for Epidemiological Studies Depression.
  It is a short self-report scale designed to measure current level of depressive symptomatology, with emphasis on the affective component, depressed mood.
  Scoring: It has 20 items each scored from 0 (Rarely or at any moment, less than a day) to 3 (Most of the time, 5-7 days).
Social isolation | Participants will be evaluated at baseline (pre-intervention), at the end of the school year (post-intervention) and at follow-up (nine months after post-intervention)
  The Social isolation questionnaire is composed of 17 items that can be categorised into three domain: feelings of loneliness, friendships, and family support.
  Scoring: The score can assume values from 0 to 117, with lower scores indicating lower levels of social isolation.
Sleep Quality | Participants will be evaluated at baseline (pre-intervention), at the end of the school year (post-intervention) and at follow-up (nine months after post-intervention)
  Sleep quality will be evaluated throught the Pittsburgh Sleep Quality Index (PSQI) questionnaire. It is a self-reported questionnaire with 19 questions grouped into 10 items.
  Scoring: In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21).

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Antunes Lima, PhD, Principal Investigator — Fundació Sant Joan de Déu
Locations (1):
- Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
This information will be used by the Research Group in charge of the investigation/s (in particular, the study researcher and his collaborators, health authorities, the promoter's monitors and auditors) who will be subject to the duty of secrecy inherent in his profession, to verify the data and procedures of the study, but always maintaining confidentiality in accordance with current legislation.
  For transfers to third countries, only encoded data will be transferred, which will in no case contain information that can directly identify you. Should this transfer occur, it would be for the same purposes described in this document and guaranteeing confidentiality. If a transfer of coded data is made outside the European Economic Area, either to entities related to the center where you participate, to service providers to researchers who collaborate with us, your data will be protected by safeguards such as contracts or other mechanisms established by data protection authorities.

REFERENCES:
- [Background] Kraft R, Hofmann F, Reichert M, Pryss R. Dealing With Inaccurate Sensor Data in the Context of Mobile Crowdsensing and mHealth. IEEE J Biomed Health Inform. 2022 Nov;26(11):5439-5449. doi: 10.1109/JBHI.2022.3198254. Epub 2022 Nov 10. PMID 35951560
- [Background] Reis RS, Salvo D, Ogilvie D, Lambert EV, Goenka S, Brownson RC; Lancet Physical Activity Series 2 Executive Committee. Scaling up physical activity interventions worldwide: stepping up to larger and smarter approaches to get people moving. Lancet. 2016 Sep 24;388(10051):1337-48. doi: 10.1016/S0140-6736(16)30728-0. Epub 2016 Jul 28. PMID 27475273
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Lee WJ, Peng LN, Lin CH, Chen RC, Lin SZ, Loh CH, Kao SL, Hung TS, Chang CY, Huang CF, Tang TC, Huang ST, Wen YW, Hsiao FY, Chen LK; Taiwan Integrated Geriatric Care Study Group. Effects of incorporating multidomain interventions into integrated primary care on quality of life: a randomised controlled trial. Lancet Healthy Longev. 2021 Nov;2(11):e712-e723. doi: 10.1016/S2666-7568(21)00248-8. Epub 2021 Oct 22. PMID 36098028
- [Background] Goodman R, Meltzer H, Bailey V. The Strengths and Difficulties Questionnaire: a pilot study on the validity of the self-report version. Eur Child Adolesc Psychiatry. 1998 Sep;7(3):125-30. doi: 10.1007/s007870050057. PMID 9826298
- [Background] Ringdal R, Bradley Eilertsen ME, Bjornsen HN, Espnes GA, Moksnes UK. Validation of two versions of the Warwick-Edinburgh Mental Well-Being Scale among Norwegian adolescents. Scand J Public Health. 2018 Nov;46(7):718-725. doi: 10.1177/1403494817735391. Epub 2017 Oct 10. PMID 29017402
- [Background] Bae S, Chung T, Ferreira D, Dey AK, Suffoletto B. Mobile phone sensors and supervised machine learning to identify alcohol use events in young adults: Implications for just-in-time adaptive interventions. Addict Behav. 2018 Aug;83:42-47. doi: 10.1016/j.addbeh.2017.11.039. Epub 2017 Nov 27. PMID 29217132
- [Background] Moshe I, Terhorst Y, Opoku Asare K, Sander LB, Ferreira D, Baumeister H, Mohr DC, Pulkki-Raback L. Predicting Symptoms of Depression and Anxiety Using Smartphone and Wearable Data. Front Psychiatry. 2021 Jan 28;12:625247. doi: 10.3389/fpsyt.2021.625247. eCollection 2021. PMID 33584388
- [Background] Dominguez-Berjon MF, Borrell C, Cano-Serral G, Esnaola S, Nolasco A, Pasarin MI, Ramis R, Saurina C, Escolar-Pujolar A. [Constructing a deprivation index based on census data in large Spanish cities(the MEDEA project)]. Gac Sanit. 2008 May-Jun;22(3):179-87. doi: 10.1157/13123961. Spanish. PMID 18579042
- [Background] Geissler J, Buchholz H, Meerson R, Kammerer K, Goster M, Schobel J, Ratz C, Taurines R, Pryss R, Romanos M. Smartphone-based behaviour analysis for challenging behaviour in intellectual and developmental disabilities and autism spectrum disorder - Study protocol for the ProVIA trial. Front Neurosci. 2022 Oct 13;16:984618. doi: 10.3389/fnins.2022.984618. eCollection 2022. PMID 36312036
- [Background] Vogel C, Schobel J, Schlee W, Engelke M, Pryss R. UNITI Mobile-EMI-Apps for a Large-Scale European Study on Tinnitus. Annu Int Conf IEEE Eng Med Biol Soc. 2021 Nov;2021:2358-2362. doi: 10.1109/EMBC46164.2021.9630482. PMID 34891756
- [Background] Schobel J, Pryss R, Probst T, Schlee W, Schickler M, Reichert M. Learnability of a Configurator Empowering End Users to Create Mobile Data Collection Instruments: Usability Study. JMIR Mhealth Uhealth. 2018 Jun 29;6(6):e148. doi: 10.2196/mhealth.9826. PMID 29959107
- [Background] Carducci B, Oh C, Keats EC, Roth DE, Bhutta ZA. Effect of Food Environment Interventions on Anthropometric Outcomes in School-Aged Children and Adolescents in Low- and Middle-Income Countries: A Systematic Review and Meta-Analysis. Curr Dev Nutr. 2020 May 26;4(7):nzaa098. doi: 10.1093/cdn/nzaa098. eCollection 2020 Jul. PMID 32666031
- [Background] Jacob CM, Hardy-Johnson PL, Inskip HM, Morris T, Parsons CM, Barrett M, Hanson M, Woods-Townsend K, Baird J. A systematic review and meta-analysis of school-based interventions with health education to reduce body mass index in adolescents aged 10 to 19 years. Int J Behav Nutr Phys Act. 2021 Jan 4;18(1):1. doi: 10.1186/s12966-020-01065-9. PMID 33397403
- [Background] Liu L, Villavicencio F, Yeung D, Perin J, Lopez G, Strong KL, Black RE. National, regional, and global causes of mortality in 5-19-year-olds from 2000 to 2019: a systematic analysis. Lancet Glob Health. 2022 Mar;10(3):e337-e347. doi: 10.1016/S2214-109X(21)00566-0. PMID 35180417
- [Background] Rageliene T, Aschemann-Witzel J, Gronhoj A. Efficacy of a smartphone application-based intervention for encouraging children's healthy eating in Denmark. Health Promot Int. 2022 Feb 17;37(1):daab081. doi: 10.1093/heapro/daab081. PMID 34245283
- [Background] Sutherland R, Reeves P, Campbell E, Lubans DR, Morgan PJ, Nathan N, Wolfenden L, Okely AD, Gillham K, Davies L, Wiggers J. Cost effectiveness of a multi-component school-based physical activity intervention targeting adolescents: the 'Physical Activity 4 Everyone' cluster randomized trial. Int J Behav Nutr Phys Act. 2016 Aug 22;13(1):94. doi: 10.1186/s12966-016-0418-2. PMID 27549382
- [Background] Hollis JL, Sutherland R, Campbell L, Morgan PJ, Lubans DR, Nathan N, Wolfenden L, Okely AD, Davies L, Williams A, Cohen KE, Oldmeadow C, Gillham K, Wiggers J. Effects of a 'school-based' physical activity intervention on adiposity in adolescents from economically disadvantaged communities: secondary outcomes of the 'Physical Activity 4 Everyone' RCT. Int J Obes (Lond). 2016 Oct;40(10):1486-1493. doi: 10.1038/ijo.2016.107. Epub 2016 Jun 10. PMID 27430652
- [Background] Sutherland RL, Campbell EM, Lubans DR, Morgan PJ, Nathan NK, Wolfenden L, Okely AD, Gillham KE, Hollis JL, Oldmeadow CJ, Williams AJ, Davies LJ, Wiese JS, Bisquera A, Wiggers JH. The Physical Activity 4 Everyone Cluster Randomized Trial: 2-Year Outcomes of a School Physical Activity Intervention Among Adolescents. Am J Prev Med. 2016 Aug;51(2):195-205. doi: 10.1016/j.amepre.2016.02.020. Epub 2016 Apr 18. PMID 27103495
- [Background] Sutherland R, Campbell E, McLaughlin M, Nathan N, Wolfenden L, Lubans DR, Morgan PJ, Gillham K, Oldmeadow C, Searles A, Reeves P, Williams M, Kajons N, Bailey A, Boyer J, Lecathelinais C, Davies L, McKenzie T, Hollis J, Wiggers J. Scale-up of the Physical Activity 4 Everyone (PA4E1) intervention in secondary schools: 12-month implementation outcomes from a cluster randomized controlled trial. Int J Behav Nutr Phys Act. 2020 Aug 8;17(1):100. doi: 10.1186/s12966-020-01000-y. PMID 32771011
- [Background] Charles MA, Thierry X, Lanoe JL, Bois C, Dufourg MN, Popa R, Cheminat M, Zaros C, Geay B. Cohort Profile: The French national cohort of children (ELFE): birth to 5 years. Int J Epidemiol. 2020 Apr 1;49(2):368-369j. doi: 10.1093/ije/dyz227. No abstract available. PMID 31747017
- [Background] Bryan CJ, Tipton E, Yeager DS. Behavioural science is unlikely to change the world without a heterogeneity revolution. Nat Hum Behav. 2021 Aug;5(8):980-989. doi: 10.1038/s41562-021-01143-3. Epub 2021 Jul 22. PMID 34294901
- [Background] Folch C, Gonzalez-Casals H, Colom J, Bosque-Prous M, Baron-Garcia T, Alvarez-Vargas A, Casabona J, Espelt A. Mental Well-Being during the COVID-19 Confinement among Adolescents in Catalonia: The Role of Demographic and Other COVID-Related Variables. Children (Basel). 2022 May 26;9(6):783. doi: 10.3390/children9060783. PMID 35740720
- [Background] Roges J, Bosque-Prous M, Colom J, Folch C, Baron-Garcia T, Gonzalez-Casals H, Fernandez E, Espelt A. Consumption of Alcohol, Cannabis, and Tobacco in a Cohort of Adolescents before and during COVID-19 Confinement. Int J Environ Res Public Health. 2021 Jul 24;18(15):7849. doi: 10.3390/ijerph18157849. PMID 34360141
- [Background] Codinach-Danes E, Obradors-Rial N, Gonzalez-Casals H, Bosque-Prous M, Folch C, Colom J, Espelt Hernandez A. Polydrug use of tobacco and cannabis: Relationship with self-perceived health and mood state in adolescents in Central Catalonia- DESKcohort Project. Adicciones. 2024 Mar 29;36(1):81-92. doi: 10.20882/adicciones.1716. English, Spanish. PMID 36200227
- [Background] Esquius L, Aguilar-Martinez A, Bosque-Prous M, Gonzalez-Casals H, Bach-Faig A, Colillas-Malet E, Salvador G, Espelt A. Social Inequalities in Breakfast Consumption among Adolescents in Spain: The DESKcohort Project. Nutrients. 2021 Jul 22;13(8):2500. doi: 10.3390/nu13082500. PMID 34444661
- [Background] Aguilar-Martinez A, Bosque-Prous M, Gonzalez-Casals H, Colillas-Malet E, Puigcorbe S, Esquius L, Espelt A. Social Inequalities in Changes in Diet in Adolescents during Confinement Due to COVID-19 in Spain: The DESKcohort Project. Nutrients. 2021 May 8;13(5):1577. doi: 10.3390/nu13051577. PMID 34066867
- [Background] Lima RA, de Barros MVG, Bezerra J, Dos Santos SJ, Monducci E, Rodriguez-Ayllon M, Soares FC. Universal school-based intervention targeting depressive symptoms in adolescents: A cluster randomized trial. Scand J Med Sci Sports. 2022 Mar;32(3):622-631. doi: 10.1111/sms.14115. Epub 2021 Dec 23. PMID 34923679
- [Background] Allgaier J, Schlee W, Probst T, Pryss R. Prediction of Tinnitus Perception Based on Daily Life MHealth Data Using Country Origin and Season. J Clin Med. 2022 Jul 22;11(15):4270. doi: 10.3390/jcm11154270. PMID 35893370
- [Background] Engelke M, Simoes J, Vogel C, Schoisswohl S, Schecklmann M, Wolflick S, Pryss R, Probst T, Langguth B, Schlee W. Pilot study of a smartphone-based tinnitus therapy using structured counseling and sound therapy: A multiple-baseline design with ecological momentary assessment. PLOS Digit Health. 2023 Jan 18;2(1):e0000183. doi: 10.1371/journal.pdig.0000183. eCollection 2023 Jan. PMID 36812641
- [Background] Baumeister H, Bauereiss N, Zarski AC, Braun L, Buntrock C, Hoherz C, Idrees AR, Kraft R, Meyer P, Nguyen TBD, Pryss R, Reichert M, Sextl T, Steinhoff M, Stenzel L, Steubl L, Terhorst Y, Titzler I, Ebert DD. Clinical and Cost-Effectiveness of PSYCHOnlineTHERAPY: Study Protocol of a Multicenter Blended Outpatient Psychotherapy Cluster Randomized Controlled Trial for Patients With Depressive and Anxiety Disorders. Front Psychiatry. 2021 May 14;12:660534. doi: 10.3389/fpsyt.2021.660534. eCollection 2021. PMID 34054617
- [Background] Lubans DR, Morgan PJ, Callister R, Collins CE. Effects of integrating pedometers, parental materials, and E-mail support within an extracurricular school sport intervention. J Adolesc Health. 2009 Feb;44(2):176-183. doi: 10.1016/j.jadohealth.2008.06.020. Epub 2008 Oct 29. PMID 19167667
- [Background] Lonsdale C, Sanders T, Parker P, Noetel M, Hartwig T, Vasconcellos D, Lee J, Antczak D, Kirwan M, Morgan P, Salmon J, Moodie M, McKay H, Bennie A, Plotnikoff RC, Cinelli R, Greene D, Peralta L, Cliff D, Kolt G, Gore J, Gao L, Boyer J, Morrison R, Hillman C, Shigeta TT, Tan E, Lubans DR. Effect of a Scalable School-Based Intervention on Cardiorespiratory Fitness in Children: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2021 Jul 1;175(7):680-688. doi: 10.1001/jamapediatrics.2021.0417. PMID 33938946
- [Background] Hartwig TB, Del Pozo-Cruz B, White RL, Sanders T, Kirwan M, Parker PD, Vasconcellos D, Lee J, Owen KB, Antczak D, Lubans DR, Lonsdale C. A monitoring system to provide feedback on student physical activity during physical education lessons. Scand J Med Sci Sports. 2019 Sep;29(9):1305-1312. doi: 10.1111/sms.13438. Epub 2019 May 23. PMID 31033042
- [Background] Smith JJ, Morgan PJ, Plotnikoff RC, Dally KA, Salmon J, Okely AD, Finn TL, Lubans DR. Smart-phone obesity prevention trial for adolescent boys in low-income communities: the ATLAS RCT. Pediatrics. 2014 Sep;134(3):e723-31. doi: 10.1542/peds.2014-1012. PMID 25157000
- [Background] Lubans DR, Smith JJ, Eather N, Leahy AA, Morgan PJ, Lonsdale C, Plotnikoff RC, Nilsson M, Kennedy SG, Holliday EG, Weaver N, Noetel M, Shigeta TT, Mavilidi MF, Valkenborghs SR, Gyawali P, Walker FR, Costigan SA, Hillman CH. Time-efficient intervention to improve older adolescents' cardiorespiratory fitness: findings from the 'Burn 2 Learn' cluster randomised controlled trial. Br J Sports Med. 2020 Dec 21;55(13):751-8. doi: 10.1136/bjsports-2020-103277. Online ahead of print. PMID 33355155
- [Background] Norris SA, Frongillo EA, Black MM, Dong Y, Fall C, Lampl M, Liese AD, Naguib M, Prentice A, Rochat T, Stephensen CB, Tinago CB, Ward KA, Wrottesley SV, Patton GC. Nutrition in adolescent growth and development. Lancet. 2022 Jan 8;399(10320):172-184. doi: 10.1016/S0140-6736(21)01590-7. Epub 2021 Nov 29. PMID 34856190
- [Background] Patton GC, Olsson CA, Skirbekk V, Saffery R, Wlodek ME, Azzopardi PS, Stonawski M, Rasmussen B, Spry E, Francis K, Bhutta ZA, Kassebaum NJ, Mokdad AH, Murray CJL, Prentice AM, Reavley N, Sheehan P, Sweeny K, Viner RM, Sawyer SM. Adolescence and the next generation. Nature. 2018 Feb 21;554(7693):458-466. doi: 10.1038/nature25759. PMID 29469095
- [Background] van Sluijs EMF, Ekelund U, Crochemore-Silva I, Guthold R, Ha A, Lubans D, Oyeyemi AL, Ding D, Katzmarzyk PT. Physical activity behaviours in adolescence: current evidence and opportunities for intervention. Lancet. 2021 Jul 31;398(10298):429-442. doi: 10.1016/S0140-6736(21)01259-9. Epub 2021 Jul 21. PMID 34302767
- [Background] Stevens K. Valuation of the Child Health Utility 9D Index. Pharmacoeconomics. 2012 Aug 1;30(8):729-47. doi: 10.2165/11599120-000000000-00000. PMID 22788262
- [Background] Lopez MA, Gabilondo A, Codony M, Garcia-Forero C, Vilagut G, Castellvi P, Ferrer M, Alonso J. Adaptation into Spanish of the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) and preliminary validation in a student sample. Qual Life Res. 2013 Jun;22(5):1099-104. doi: 10.1007/s11136-012-0238-z. Epub 2012 Jul 27. PMID 22836376
- [Background] Ravens-Sieberer U, Gosch A, Rajmil L, Erhart M, Bruil J, Duer W, Auquier P, Power M, Abel T, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J, Kidscreen Group E. KIDSCREEN-52 quality-of-life measure for children and adolescents. Expert Rev Pharmacoecon Outcomes Res. 2005 Jun;5(3):353-64. doi: 10.1586/14737167.5.3.353. PMID 19807604
- [Background] Johnson F, Wardle J, Griffith J. The Adolescent Food Habits Checklist: reliability and validity of a measure of healthy eating behaviour in adolescents. Eur J Clin Nutr. 2002 Jul;56(7):644-9. doi: 10.1038/sj.ejcn.1601371. PMID 12080404

DOCUMENTS (1):
  • Informed Consent Form (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT06792461/ICF_000.pdf